CLINICAL TRIAL: NCT00992914
Title: Pilot Study of Stellate Ganglion Injection With Anesthetic as a Method to Provide Relief From Hot Flushes
Brief Title: Pilot Study of Stellate Ganglion Injection to Provide Relief From Hot Flushes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Lee Shulman, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU6644
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Hot Flashes; Menopause
Keywords: Hot flushes (vasomotor symptoms)
MeSH Terms: conditions — Hot Flashes | interventions — Autonomic Nerve Block; Lidocaine

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine injection (Active Comparator): Stellate Ganglion Injection with Lidocaine
  Interventions: Procedure: Sympathetic nerve block with 1% lidocaine 1-2 ml
- saline injection (Placebo Comparator): Superficial subcutaneous injection
  Interventions: Procedure: Superficial subcutaneous injection

INTERVENTIONS:
Procedure: Sympathetic nerve block with 1% lidocaine 1-2 ml — Stellate Ganglion Injection
  Arms: Lidocaine injection
Procedure: Superficial subcutaneous injection — Superficial subcutaneous injection with saline
  Arms: saline injection

SUMMARY:
This study is being done to determine whether stellate ganglion injection with local anesthetic (the study procedure) can reduce the number and severity of hot flashes in women who have hot flashes.

Hot flashes can have a significant impact on daily living, disrupt sleep, and lead to fatigue and irritability during the day. Hot flashes are the most common reason that women seek hormonal therapy. However, for many women, including breast cancer survivors, this is rarely an option, and these women seek alternatives to hormonal therapy to treat hot flashes.

The study procedure has been in clinical use for more than fifty years in treating certain disease states and chronic pain. The study procedure has not been used to relieve hot flashes and the use of the study procedure with local anesthetic for the reduction of hot flushes is considered experimental.

ELIGIBILITY:
Inclusion Criteria:

* Women surgically or naturally menopausal,
* Experiencing moderate to severe hot flushes, AND
* Elect to undergo stellate ganglion block procedure.

Exclusion Criteria:

* Subjects who are currently sick,
* Subjects have acute infections or cardiac compromise,
* Subjects who have local infections of the anterior neck region, severe
* Subjects who have pulmonary disease,
* Subjects who are anticoagulated,
* Subjects who are on hormone therapy,
* Subjects who have a blood clotting disorder,
* Subjects who have an American Society of Anesthesiologists (ASA) physical status score of 3 or higher (severe systemic disease, not incapacitating),
* Subjects who have allergic reactions to local anesthetics and/or contrast dyes,
* Subjects who have past or present diagnosis of psychosis,
* Subjects who have current diagnosis of depression, OR
* Subjects who have current substance or alcohol abuse.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-02; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Reduction of hot flushes. | 6 months

SECONDARY OUTCOMES:
To investigate the impact of stellate ganglion injection with local anesthetic on cognitive function. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lee P Shulman, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States